CLINICAL TRIAL: NCT02156791
Title: Safety, Clinical Tolerability and Immunogenicity of Increasing Doses of gpASIT+TM Administered Subcutaneously to Hay Fever Patients
Brief Title: Safety, Clinical Tolerability and Immunogenicity of Increasing Doses of gpASIT+TM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioTech Tools S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTT-gpASIT007
Record Dates: First submitted 2014-05-23; First posted 2014-06-05 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-05

CONDITIONS: Hay Fever
Keywords: Seasonal allergic rhinoconjunctivitis; Grass pollen; Allergen specific immunotherapy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- gpASIT+TM (Experimental)
  Interventions: Biological: gpASIT+TM

INTERVENTIONS:
Biological: gpASIT+TM

SUMMARY:
gpASIT+TM product is based on highly purified allergen fragments obtained from grass pollen. The purpose of this clinical trial is to confirm the safety, clinical tolerability and immunogenicity of increasing doses of gpASIT+TM administered subcutaneously to patients with grass pollen-induced allergic rhinoconjunctivitis, and to determine the maximal tolerated dose of gpASIT+TM .

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated Informed Consent Form by a legally competent patient
* Female or male patients aged 18-70 years
* The patients are in good physical and mental health according to his/her medical history and vital signs
* Non-pregnant, non-lactating females with adequate contraception
* Females unable to bear children must have signed the form for adequate contraceptive protection (i.e. tubule ligation, hysterectomy, or post-menopausal (defined as a minimum of one year since the last menstrual period))
* Allergy diagnosis:

  * A medical history of moderate to severe seasonal allergic rhinoconjunctivitis (SAR) for the grass pollen season during at least the two previous years
  * A positive skin prick test (wheal diameter ≥ 3 mm) to grass-pollen mixture, histamine wheal ≥ 3 mm, NaCl control reaction ≤ 2 mm
  * Specific IgE against grass pollen (IgE > 0.7 kU/l)
  * Patients treated with anti-allergic medication for at least 2 years prior to enrolment
* In asthmatic patients:

  * Confirmed diagnosis of controlled asthma according to GINA-guidelines (GINA 2011)

Exclusion Criteria:

* Simultaneous participation in other clinical trials or previous participation within 30 days before inclusion
* Previous immunotherapy with grass allergens within the last 5 years
* Ongoing immunotherapy
* Patients being in any relationship or dependence with the Sponsor and/ or Investigator
* Inability to understand instructions/ study documents
* Patients with a history of hypersensitivity to the excipients of investigational products
* Patients with partly controlled or uncontrolled asthma
* Chronic asthma or emphysema, particularly with a FEV 1 <80% of the predicted value (ECSC)
* Patients symptomatic to perennial inhalant allergens to which the subjects are regularly exposed
* Patients with a history of ragweed allergy
* Patients with a history of renal disease or chronic hepatic disease
* Patients with malignant disease
* Patients with a know severe autoimmune disease and patients with a positive test to ANA, ANCA or ASCA
* Patients with any chronic disease which may impair the patient's ability to participate in the trial (i.e. severe congestive heart failure, active gastric ulcer, inflammatory bowel disease, uncontrolled diabetes mellitus, etc…)
* Patients requiring beta-blockers/ACE-inhibitors medication
* Patients requiring anti-IgE antibodies, mast cell stabilizers, and antileukotriene agents
* Patients with any contraindication for the use of adrenaline
* Patients with febrile illness (> 37.5°C, oral)
* Patients with a known positive serology for HIV-1/2, HBV or HCV
* Patients who are immunocompromised by medication or illness, have received a vaccine corticoids or immunosuppressive medications within 1 month before trial entry
* Female patients who are pregnant, lactating, or of child-bearing potential and not protected from pregnancy by a sufficiently reliable method
* Consumption of corticoids (oral, topic or nasal) or of anti-histaminic drugs within 3 weeks preceding the trial (screening visit)
* Patients with laboratory values greater than grade 1 according to the FDA Guidance for Industry for preventive Vaccine Trials (FDA 2007)
* Unreliable patients including non-compliant patients, patients with known alcoholism or drug abuse or with a history of a serious psychiatric disorder as well as patients unwilling to give informed consent or to abide by the requirements of the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
(Serious) adverse events | Up to 6 weeks

SECONDARY OUTCOMES:
Grass pollen allergen -specific immunoglobulins | up to 6 weeks
Blocking antibody production | up to 6 weeks
Change from baseline in Conjunctival Provocation Test score | at screening, after 4 weeks and 6 weeks of treatment
Local reaction at the injection site | up to 6 weeks
Systemic reaction after injection | up to 6 weeks
Change from baseline in safety laboratory parameters | up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Hauswald, MD, Principal Investigator — Universitätsklinikum Carl-Gustav-Carus, Dresden, Germany
Locations (1):
- Universitätsklinikum Carl-Gustav-Carus, Dresden, Germany, Dresden, Germany